CLINICAL TRIAL: NCT03713788
Title: Muscle Stretching - the Potential Role of Endogenous Pain Inhibitory Modulation on Stretch Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Northern Denmark (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Morten Pallisgaard, Senior associate lecturer, University College of Northern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UniversityCND
Record Dates: First submitted 2018-10-15; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Muscle Stretching Exercises; Pain Threshold
Keywords: Stretch tolerance; Range of Motion

STUDY DESIGN:
Intervention Model Description: A sample of convenience was recruited for this cross-sectional study. Participants were randomly assigned to a pain group or a control group using counterbalanced block randomization. Passive knee extension range of motion was measured three consecutive times with five-minute intervals between measurements. Both groups underwent a static stretch protocol consisting of two bouts of thirty-second constant-angle static stretching of the knee flexors with a one-minute rest between bouts. Subjects were instructed to keep the limb relaxed as the lower leg was passively moved towards extension. Following stretching, the post-stretch measurement was performed. Finally, subjects in the pain group were instructed to immerse their non-dominant hand into a container with circulating water at 1˚C to 4˚C and keep it there for 2 minutes. A Biodex system 4 pro dynamometer was used to quantify range of motion and passive resistive torque. Muscle activity was recorded as surface electromyography.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental pain group (Experimental): subjects in the pain group were instructed to immerse their non-dominant hand into a container with circulating water at 1˚C to 4˚C and keep it there for 2 minutes. They were instructed to immerse it to wrist-level and keep the hand open.
  Interventions: Other: Cold pressor test
- Control group (No Intervention): Participants rested in a seated position for 5 minutes.

INTERVENTIONS:
Other: Cold pressor test — Participants placed their non-dominant hand into cold water for 2 minutes
  Arms: Experimental pain group

SUMMARY:
This study investigates the influence of a remote, painful stimulus on stretch tolerance. Half of the participants will receive a conditioning painful stimulus following static stretching while the other half will rest quietly.

DETAILED DESCRIPTION:
The effect of stretching on joint range of motion is primarily related to changes in the tolerance to stretch, but the mechanisms underlying this change are still largely unknown.

The nervous system has an inbuilt ability to modulate the perceived magnitude of afferent noxious stimuli via supraspinally mediated endogenous pain inhibition or facilitation and by engaging endogenous mechanisms pain tolerance in healthy individuals is known to increase. Thus increasing the tolerance to pain could potentially increase range of motion following stretching.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for participation included the absence of any pain or other conditions that might affect the somatosensory system.

Exclusion Criteria:

* Substance abuse,
* History of neurological or mental disabilities
* Lack of ability to comply with instructions
* Delayed onset of muscle soreness.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only males were included to avoid the potential effect that fluctuations in gonadal hormone values may have on the endogenous pain inhibitory mechanisms.
Enrollment: 34 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Knee extension range of motion | Passive knee extension range of motion was measured at baseline
  Passively induced knee extension range of motion was measured usind the Biodex system 4 pro isokinetic dynomometer
Change in knee extension range of motion between baseline and post stretch. | Changes in passive knee extension range of motion were measured 5 minutes after baseline measures following stretching
  Changes in passively induced knee extension range of motion was measured using the Biodex system 4 pro isokinetic dynomometer
Changes in knee extension range of motion between post stretch and post pain. | Changes in passive knee extension range of motion were measured 5 minutes after post stretch measures following intervention.
  Changes in passively induced knee extension range of motion was measured using the Biodex system 4 pro isokinetic dynomometer

SECONDARY OUTCOMES:
Surface electromyography measures of muscle activity | Muscle activity during the passive knee extension motion was measured at baseline
  Muscle activity during the passive knee extension motion were measured using SEMG.
Changes in surface electromyography measures of muscle activity between baseline and post stretch measures. | Changes in muscle activity during the passive knee extension motion were measured 5 minutes after baseline measures following stretching.
  Changes in muscle activity during the passive knee extension motion were measured using SEMG.
Changes in surface electromyography measures of muscle activity between post stretch and post pain measures. | Changes in muscle activity during the passive knee extension motion were measured 5 minutes after post stretch measures following intervention.
  Changes in muscle activity during the passive knee extension motion were measured using SEMG.
Passive resistive torque using the Biodes system 4 pro. | Passive resistive torque during the passive knee extension motion was measured at baseline.
  Passive resistive torque during the passive knee extension motion was measured using the Biodex system 4 pro isokinetic dynamometer.
Changes in passive resistive torque measured using the Biodex system 4 pro between baseline and post stretch measures. | Changes in passive resistive torque during the passive knee extension motion was measured 5 minutes after baseline measures following stretching.
  Changes in passive resistive torque during the passive knee extension motion was measured using the Biodex system 4 pro isokinetic dynamometer.
Changes in passive resistive torque measured using the Biodex system 4 pro between post stretch and post pain measures. | Passive resistive torque during the passive knee extension motion was measured 5 minutes after post stretch measures following intervention.
  Changes in Passive resistive torque during the passive knee extension motion was measured using the Biodex system 4 pro isokinetic dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Drachman, Msc., Study Director — University College of Northern Denmark, Department of Physiotherapy
Locations (1):
- University College of Northern Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No